CLINICAL TRIAL: NCT01357915
Title: A Follow-up Study to Evaluate the Long-term Persistence of GSK Biologicals' Candidate CMV Vaccine Administered to Male Adults
Brief Title: Evaluation of the Long-term Persistence of GlaxoSmithKline (GSK) Biologicals' Candidate Cytomegalovirus (CMV) Vaccine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 115429; 2011-002702-78 (EudraCT Number)
Record Dates: First submitted 2011-05-12; First posted 2011-05-23 (Estimated); Results first posted 2017-10-06 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Infections, Cytomegalovirus
Keywords: Cytomegalovirus; Vaccine
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Blood Specimen Collection

ARMS (2):
- GSK149203A S- Group (Experimental): Male subjects who received 3 doses of GSK Biologicals' candidate GSK149203A vaccine according to a 0-1-6 month schedule in the primary study 108890 (NCT00435396).
  Interventions: Procedure: Blood sampling; Biological: GSK149203A
- GSK149203A S+ Group (Other): Male subjects who were assessed as being naturally infected with Cytomegalovirus (CMV) at the screening visit of the primary study 108890 (NCT00435396).
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — Blood samples will be collected at 2 time points:
  At the long-term follow-up at approximately Month 48 of study (= ± 42 months post dose 3) from all subjects in the vaccine group.
  At the long-term follow-up at approximately Month 60 of study (= ± 54 months post dose 3) from all subjects.
Biological: GSK149203A — GSK Biologicals' Recombinant CMV glycoprotein B Vaccine, Intramuscular injection, 3 doses
  Arms: GSK149203A S- Group

SUMMARY:
The purpose of this study is to evaluate the persistence of the vaccine induced immune responses at Month 48 (Year 4) and Month 60 (Year 5) in healthy subjects who received 3 doses of GSK Biologicals' candidate CMV vaccine according to a 0-1-6 month schedule during the primary study 108890 (NCT00435396) (vaccine group). The immune response to CMV infection in naturally infected subjects who participated in the screening visit of the primary study 108890 (NCT00435396) and who were tested CMV-seropositive, will be used as a reference value (seropositive reference group). In addition, this study will continue to assess the occurrence of CMV infections as well as the continued development and validation of read-outs in the CMV project.

The primary vaccination phase and Year 2 follow-up were posted as a separate protocol posting (NCT00435396).

DETAILED DESCRIPTION:
During the long-term follow-up study, all subjects who received 3 doses of GSK Biologicals' candidate CMV vaccine according to a 0-1-6 month schedule during the primary study 108890 (NCT00435396) will be invited to participate at Visit 8 (Year 4) and Visit 9 (Year 5) as the vaccine group. In addition, the healthy subjects who participated in the screening visit of the primary study 108890 (NCT00435396) and who were tested CMV-seropositive will be invited to Visit 9 (Year 5) of this study as the seropositive reference group.This Protocol Posting has been updated following Protocol Amendment 1, March 2012, leading to the update of brief summary, intervention model, enrolment, outcome measures, eligibility and arms.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol (e.g., return for follow-up visits) should be enrolled in the study.
* Written informed consent obtained from the subject.
* Healthy subjects as established by clinical evaluation (medical history and physical examination) before entering in the study.

Subjects of the vaccine group should in addition satisfy the following criterion:

• Subjects who participated in the primary study 108890 (NCT00435396), having received 3 doses of the GSK's CMV candidate vaccine and having completed the Year 2 follow-up study 109211 (NCT00435396).

Subjects of the seropositive reference group should in addition satisfy the following criterion:

• Subjects who participated in the screening visit of the primary study 108890 (NCT00435396), and whose blood sample taken at this visit was tested CMV positive.

Exclusion Criteria:

* Use, or planned use, of any investigational or non-registered product (drug or vaccine) during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to study visit(s). For corticosteroids, this will mean prednisone, 20mg/day, or equivalent. Inhaled and topical steroids are allowed.
* Administration of immunoglobulins and/or any blood products within three months preceding study visit(s).
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).

For subjects in the vaccine group, the following exclusion criterion should be checked in addition:

• Administration of any additional CMV vaccine since end of primary study 108890 (NCT00435396).

For subjects in the seropositive reference group, the following exclusion criterion should be checked in addition:

• Administration of any CMV vaccine since the screening visit of primary study 108890 (NCT00435396).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2011-06-24 (Actual); Primary Completion 2012-09-13 (Actual); Study Completion 2012-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Belgium (2):
  - GSK Investigational Site, La Louvière
  - GSK Investigational Site, Wilrijk

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects from the GSK149203A S+ Group participated only in the Month 60 time point of the study.
Groups:
- GSK149203A S- Group: Healthy male subjects who received 3 doses of GSK Biologicals' candidate GSK149203A vaccine according to a 0-1-6 month schedule in the primary study 108890 (NCT00435396).
- GSK149203A S+ Group: Healthy male subjects who were assessed as being naturally infected with Cytomegalovirus (CMV) at the screening visit of the primary study 108890 (NCT00435396).
Period: Overall Study
Arm/Group | GSK149203A S- Group | GSK149203A S+ Group
Started | 30 | 17
Completed | 27 | 17
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK149203A S- Group | GSK149203A S+ Group | Total
Number analyzed (Participants) | 30 | 17 | 47
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.3 (6.37) | 35.5 (7.20) | 34.73 (6.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 30 | 17 | 47
Race/Ethnicity, Customized [Number; unit: Participants]
  White-Caucasian/European heritage | 30 | 16 | 46
  Other: unknown | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Concentrations of Antibodies Against Anti-Glycoprotein B (gB) Immunoglobulin G (IgG)
Description: Anti-gB IgG antibody concentrations were presented as Geometric Mean Concentrations (GMCs) and expressed in ELISA units per milliliter (EL.U/mL), as assessed by Enzyme-linked Immunosorbent Assay (ELISA). Data were collected at Month 48 (M48) and Month 60 (M60) from all subjects.
Time Frame: At Month 48 and Month 60
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK149203A S- Group | GSK149203A S+ Group
Number analyzed (Participants) | 27 | 16
EL.U/mL
  Anti-gB IgG, M48: number analyzed (Participants) | 27 | 0
  Anti-gB IgG, M48 | 5091.4 [3463.2 to 7485.1] |
  Anti-gB IgG, M60 | 5495.1 [3594.7 to 8400.1] | 2587.2 [1745.6 to 3834.5]

2. Primary Outcome: Number of Subjects With Neutralizing Response Against Anti-Cytomegalovirus (CMV) Antibodies
Description: The neutralizing antibodies were to be measured using an in-house micro-neutralization assay.
Time Frame: At Month 48 and Month 60
Population: The persistence of the functional antibodies for Month 48 and Month 60 could not be analysed, due to the general deterioration of CMV-001/CMV-008 samples.
Arm/Group | GSK149203A S- Group | GSK149203A S+ Group
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Descriptive Statistics on Avidity Index (%) of Anti-gB IgG Antibodies
Description: Avidity for anti-gB IgG antibodies was assessed by the ELISA Avidity index method in all subjects, at Month 48 (M48) and Month 60 (M60).
  This assay has been developed according to Souza et al (Rev.Inst.med.Trop.S.Paulo 45;323-326; 2003) using an elution step with urea to remove low-avidity antibodies from CMV antigen. The avidity index was calculated as the mean absorbance of reactions in which the immune complexes are exposed to urea divided by the mean absorbance of reactions in which the immune complexes are not exposed to urea, expressed as a percentage.
Time Frame: At Month 48 and Month 60
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available.
Measure: Median (Inter-Quartile Range); unit: Avidity Index percentage
Arm/Group | GSK149203A S- Group | GSK149203A S+ Group
Number analyzed (Participants) | 27 | 16
Avidity Index percentage
  Anti-gB IgG, M48: number analyzed (Participants) | 27 | 0
  Anti-gB IgG, M48 | 74 [70 to 76] |
  Anti-gB IgG, M60 | 68 [65 to 71] | 76 [71.5 to 82.5]

4. Secondary Outcome: Descriptive Statistics on the Frequency of gB-specific Cluster of Differentiation (CD4+/CD8+) T-cells Expressing at Least Two Immune Markers
Description: Among the immune markers determined by the Intracellular cytokine staining (ICS) were Interferon-gamma (INF-γ), Interleukin-2 (IL-2), Tumor necrosis factor-alpha (TNF-α), and CD40-Ligand (CD40-L). Data were collected for all subjects at Month 48 (M48) and Month 60 (M60).
Time Frame: At Month 48 and Month 60
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK149203A S- Group | GSK149203A S+ Group
Number analyzed (Participants) | 26 | 15
T cells/million cells
  CD4-All doubles, M48: number analyzed (Participants) | 25 | 0
  CD4-All doubles, M48 | 2169.00 [1391.00 to 4290.00] |
  CD4-All doubles, M60 | 1893.50 [1070.00 to 3267.00] | 380.00 [91.00 to 1704.00]
  CD8-All doubles, M48: number analyzed (Participants) | 25 | 0
  CD8-All doubles, M48 | 91.00 [1.00 to 173.00] |
  CD8-All doubles, M60 | 104.00 [24.00 to 287.00] | 81.00 [2.00 to 321.00]

5. Secondary Outcome: Desciptive Statistics on the Frequency of gB-specific Memory B-cells (by ELISPOT)
Description: Memory B cells specific to the CMV gB antigen, as assessed by the Enzyme-linked Immunosorbent Spot (ELISPOT) method, were expressed as a frequency of the specific memory B-cells per million memory B-cells. Data were collected for all subjects at Month 48 (M48) and Month 60 (M60).
Time Frame: At Month 48 and Month 60
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: B cells/million cells
Arm/Group | GSK149203A S- Group | GSK149203A S+ Group
Number analyzed (Participants) | 27 | 16
B cells/million cells
  Memory B-cells, M48: number analyzed (Participants) | 27 | 0
  Memory B-cells, M48 | 3158.00 [1467.00 to 7419.00] |
  Memory B-cells, M60: number analyzed (Participants) | 26 | 16
  Memory B-cells, M60 | 5784.00 [4374.00 to 7240.00] | 210.50 [46.00 to 676.50]

6. Secondary Outcome: Number of Subjects With Response for Anti-CMV Tegument IgG Antibodies
Description: CMV infection was determined by the anti-CMV proteins antibody response, using ELISA. Data were collected for all subjects at Month 48 (M48) and Month 60 (M60) in the Vaccine group (GSK149203A S- Group). All subjects from the Reference group (GSK149203A S+ Group) were positive for the anti-CMV tegument IgG antibodies at the screening visit.
Time Frame: At Month 48 and Month 60
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK149203A S- Group
Number analyzed (Participants) | 30
Participants
  Positive anti-CMV antibodies, M48 | 0
  Negative anti-CMV antibodies, M48 | 26
  Missing anti-CMV antibodies, M48 | 4
  Positive anti-CMV antibodies, M60 | 2
  Negative anti-CMV antibodies, M60 | 25
  Missing anti-CMV antibodies, M60 | 3

7. Secondary Outcome: Assessment of CMV Infection by CMV Specific Desoxyribonucleic Acid (DNA) in Viral Load
Description: CMV DNA viral loads were assessed using quantitative Polymerase Chain Reaction (qPCR). Data were presented for subjects included in the Vaccine group (GSK149203A S- Group).
Time Frame: At Month 48 and Month 60
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK149203A S- Group
Number analyzed (Participants) | 30
Participants | NA — In the vaccine group, at Month 48 and Month 60 after the first vaccination, none of the subjects assessed had CMV DNA detected in blood (by qPCR), the values were under 200.

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (SAEs) and other adverse events: during the entire study period (from Month 48 up to Month 60) there were no SAEs or other significant AEs reported in the study.
Description: Other (non-serious) Adverse Events were not collected in the study.
Arm/Group | GSK149203A S- Group | GSK149203A S+ Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/17
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.